CLINICAL TRIAL: NCT04386746
Title: A Phase II Trial for the Use of Intravesical Gemcitabine and Docetaxel (GEMDOCE) in the Treatment of BCG naïve Non-muscle Invasive Urothelial Carcinoma of the Bladder
Brief Title: Intravesical Gemcitabine and Docetaxel for BCG naïve Non-muscle Invasive Bladder Cancer
Acronym: GEMDOCE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2020; IRB00241941 (Other: Johns Hopkins Institutional Review Boards)
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Urothelial Carcinoma Bladder; Bladder Cancer
Keywords: NMIBC
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intravesical Gemcitabine/Docetaxel (Experimental): Gemcitabine/Docetaxel induction is given intravesically in sequential order once a week for six consecutive weeks. One gram of gemcitabine in 50 ml of sterile water is slowly instilled into the bladder via a Foley catheter and the catheter is clamped for 60 minutes. The bladder is then drained and 40 mg of docetaxel in 50 ml of NSS is then slowly instilled via the Foley catheter into the bladder. The catheter is again clamped for 60 minutes before draining. If initial efficacy seen, patients will have monthly maintenance instillations of Gemcitabine/Docetaxel.
  Interventions: Drug: Gemcitabine; Drug: Docetaxel

INTERVENTIONS:
Drug: Gemcitabine — 1g gemcitabine in 50ml sterile water; instilled once weekly for 6 weeks and then once monthly for ≤ 21 months.
  Other Names: Gemzar
Drug: Docetaxel — 37.5mg docetaxel in 50ml normal saline solution (NSS); instilled once weekly for 6 weeks and then once monthly for ≤ 21 months.
  Other Names: Taxotere

SUMMARY:
A single-arm, two-stage, open-label, phase 2 study investigating the safety and efficacy of intravesical gemcitabine/docetaxel for bacillus Calmette-Guerin (BCG)-naïve patients with non-muscle invasive bladder cancer (NMIBC).

DETAILED DESCRIPTION:
All participants will receive an induction course of gemcitabine/docetaxel instillations (administered once a week for six consecutive weeks) followed by monthly maintenance instillations if initial efficacy is seen. In addition to providing initial efficacy data, this study will provide safety and long-term efficacy data on the combination regimen studied. A tolerable safety profile and demonstrated efficacy would support a potential, randomized phase 3 trial comparing the experimental combination therapy and standard of care intravesical BCG therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed intermediate or high-risk non-muscle invasive urothelial carcinoma of the bladder (Ta, T1, or Tis stage) on TURBT obtained within 90 days of registration defined according to modified EORTC risk criteria summarized as follows:

   1. Low-risk tumors: Initial or recurrent tumor > 12 months after resection with all of the following:

      * Solitary tumor
      * Low-grade
      * < 3 cm
      * No carcinoma in situ (CIS)
   2. Intermediate-risk tumors: All tumors not defined in the two adjacent categories (between the category of low- and high-risk)
   3. High-risk tumors: Any of the following:

      * T1 tumor
      * High-grade
      * CIS
      * Multiple and recurrent and large (> 3 cm) Ta low-grade tumors (all conditions must be met for this point of Ta low-grade tumors)
   4. Note #1: Low-risk tumors as defined above are not eligible
   5. Note #2: Mixed histologies are permitted, provided a component of urothelial carcinoma is present
   6. Note #3: All patients with high-grade T1 (HGT1) should undergo a restaging TURBT
2. Eastern Cooperative Oncology Group (ECOG) (WHO) performance status 0, 1, or 2
3. Age ≥ 18 years old at time of consent
4. Evidence of post-menopausal status or negative urinary or serum pregnancy test or female pre-menopausal patients is required. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   1. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
5. Subjects who give a written informed consent obtained according to local guidelines.

Exclusion Criteria:

1. Subjects with muscle-invasive (i.e. T2, T3, T4), locally advanced unresectable, or metastatic urothelial carcinoma as assessed on baseline radiographic imaging obtained within 90 days prior to study registration. The required radiographic imaging includes:

   1. Abdomen/Pelvis - CT scan
   2. Chest - chest x-ray or CT scan
2. Subjects with concurrent upper urinary tract (i.e. ureter, renal pelvis) urothelial carcinoma of any stage.

   a. Note: Subjects with history of non-invasive (Ta, Tis) upper tract urothelial carcinoma that has been definitively treated with at least one post-treatment disease assessment (i.e. cytology, biopsy, imaging) that demonstrates no evidence of residual disease are eligible.
3. Subjects with another active second malignancy with an estimated overall survival from the second malignancy of < 12 months. Subjects with another second active malignancy that are deemed to have an estimated overall survival of >12 months are eligible.
4. Subjects who have received the last administration of an anti-cancer therapy including chemotherapy, immunotherapy, and monoclonal antibodies ≤ 4 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy.
5. Subjects who have had radiotherapy ≤ 4 weeks prior to starting study drug, or who have not recovered from radiotherapy toxicities.
6. Pregnant or breast-feeding women.
7. Subjects unwilling or unable to comply with the protocol.
8. Patients with prior systemic gemcitabine or docetaxel use for a non-bladder malignancy may enroll and receive treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2026-11-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Max Kates, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University: Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sidney Kimmel Comprehensive Cancer Center website — https://www.hopkinsmedicine.org/kimmel_cancer_center/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 subjects signed consent to be screened for eligibility.
  * 1 subject signed consent, but did not meet the eligibility criteria to start the study (screen failure)
  * 26 subjects received study treatment (1 subject withdrew consent after first dose of study therapy)
Period: Overall Study
Arm/Group | Intravesical Gemcitabine/Docetaxel
Started | 26
Completed | 4
Not Completed | 22

BASELINE CHARACTERISTICS:
Arm/Group | Intravesical Gemcitabine/Docetaxel
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Pre-trial pathologic stage [Count of Participants; unit: Participants] — High-grade (HG) bladder cancer is described as more likely to grow and spread after treatment.T1 is defined as cancer that has grown into the layer of connective tissue under the lining layer of the bladder, but has not reached the layer of muscle in the bladder wall.vCIS is defined as cancer that is flat.Ta is defined as cancer that has grown toward the hollow center of the bladder but has not grown into the connective tissue or muscle of the bladder wall (non-invasive papillary carcinoma).
  Pathologic staging order of better to worse prognosis: HGTa, CIS, HGT1 without CIS, and HGT1 with CIS.
  Participants
    HGT1 with CIS | 7
    HGT1 without CIS | 7
    HgTa | 9
    CIS alone | 3

OUTCOME MEASURES:

1. Primary Outcome: 3-Month Complete Response Rate
Description: Number of patients with no evidence of recurrent high grade urothelial carcinoma of the bladder of any stage as assessed by cystoscopy with biopsy and urine cytology.
Time Frame: 3 months
Population: 1 patient withdrew consent and data was not collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravesical Gemcitabine/Docetaxel
Number analyzed (Participants) | 25
Participants | 25

2. Secondary Outcome: 12-Month Relapse-Free Survival Rate
Description: Proportion of patients alive and with no evidence of recurrent high grade urothelial carcinoma of the bladder of any stage.
Time Frame: 12 months
Reporting Status: Not Posted

3. Secondary Outcome: 24-Month Relapse-Free Survival Rate
Description: as for outcome 2
Time Frame: 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Safety Profile as Assessed by Proportion of Adverse Events by Type
Description: Proportion of adverse events by type, as defined by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Time Frame: Up to 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Safety Profile as Assessed by Proportion of Adverse Events by Grade
Description: Proportion of adverse events by grade, as defined by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Time Frame: Up to 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Number of Gene Alterations as Measured by RNA-seq
Description: Number of gene alterations as measured by RNA-seq. Compare results to 3-month Complete Response rate using statistical methods.
Time Frame: 3 months
Reporting Status: Not Posted

7. Secondary Outcome: Type of Gene Alterations as Measured by RNA-seq
Description: Type of gene alterations as measured by RNA-seq. Compare results to 3-month Complete Response rate using statistical methods.
Time Frame: 3 months
Reporting Status: Not Posted

8. Secondary Outcome: Number of Gene Alterations as Measured by RNA-seq
Description: Number of gene alterations as measured by RNA-seq. Compare results to 12-month Relapse-Free Survival rate using statistical methods.
Time Frame: 12 months
Reporting Status: Not Posted

9. Secondary Outcome: Type of Gene Alterations as Measured by RNA-seq
Description: Type of gene alterations as measured by RNA-seq. Compare results to 12-month Relapse-Free Survival rate using statistical methods.
Time Frame: 12 months
Reporting Status: Not Posted

10. Secondary Outcome: Number of DNA Mutations as Measured by Whole Transcriptome
Description: Number of DNA mutations as measured by whole transcriptome. Compare results to 3-month Complete Response rate.
Time Frame: 3 months
Reporting Status: Not Posted

11. Secondary Outcome: Number of DNA Mutations as Measured by Whole Exome
Description: Number of DNA mutations as measured by whole exome. Compare results to 3-month Complete Response rate.
Time Frame: 3 months
Reporting Status: Not Posted

12. Secondary Outcome: Number of DNA Mutations as Measured by Panel DNA Sequencing
Description: Number of DNA mutations as measured by panel DNA sequencing. Compare results to 3-month Complete Response rate.
Time Frame: 3 months
Reporting Status: Not Posted

13. Secondary Outcome: Type of DNA Mutations as Measured by Whole Transcriptome
Description: Type of DNA mutations as measured by whole transcriptome. Compare results to 3-month Complete Response rate.
Time Frame: 3 months
Reporting Status: Not Posted

14. Secondary Outcome: Type of DNA Mutations as Measured by Whole Exome
Description: Type of DNA mutations as measured by whole exome. Compare results to 3-month Complete Response rate.
Time Frame: 3 months
Reporting Status: Not Posted

15. Secondary Outcome: Type of DNA Mutations as Measured by Panel DNA Sequencing
Description: Type of DNA mutations as measured by panel DNA sequencing. Compare results to 3-month Complete Response rate.
Time Frame: 3 months
Reporting Status: Not Posted

16. Secondary Outcome: Number of DNA Mutations as Measured by Whole Transcriptome
Description: Number of DNA mutations as measured by whole transcriptome. Compare results to 12-month Relapse Free Survival rate using statistical analysis.
Time Frame: 12 months
Reporting Status: Not Posted

17. Secondary Outcome: Number of DNA Mutations as Measured by Whole Exome
Description: Number of DNA mutations as measured by whole exome. Compare results to 12-month Relapse Free Survival rate using statistical analysis.
Time Frame: 12 months
Reporting Status: Not Posted

18. Secondary Outcome: Number of DNA Mutations as Measured by Panel DNA Sequencing
Description: Number of DNA mutations as measured by panel DNA sequencing. Compare results to 12-month Relapse Free Survival rate using statistical analysis.
Time Frame: 12 months
Reporting Status: Not Posted

19. Secondary Outcome: Type of DNA Mutations as Measured by Whole Transcriptome
Description: Type of DNA mutations as measured by whole transcriptome. Compare results to 12-month Relapse Free Survival rate using statistical analysis.
Time Frame: 12 months
Reporting Status: Not Posted

20. Secondary Outcome: Type of DNA Mutations as Measured by Whole Exome
Description: Type of DNA mutations as measured by whole exome. Compare results to 12-month Relapse Free Survival rate using statistical analysis.
Time Frame: 12 months
Reporting Status: Not Posted

21. Secondary Outcome: Type of DNA Mutations as Measured by Panel DNA Sequencing
Description: Type of DNA mutations as measured by panel DNA sequencing. Compare results to 12-month Relapse Free Survival rate using statistical analysis.
Time Frame: 12 months
Reporting Status: Not Posted

22. Secondary Outcome: Numbers of T-cell Subpopulations
Description: Numbers of t-cell subpopulations utilizing immunohistochemical (IHC) staining and flow cytometry. Compare results to 3-month Complete Response rate using statistical analysis.
Time Frame: 3 months
Reporting Status: Not Posted

23. Secondary Outcome: Ratio of T-cell Subpopulations
Description: Ratio of t-cell subpopulations utilizing IHC staining and flow cytometry. Compare results to 3-month Complete Response rate using statistical analysis.
Time Frame: 3 months
Reporting Status: Not Posted

24. Secondary Outcome: Numbers of T-cell Subpopulations
Description: Numbers of t-cell subpopulations utilizing IHC staining and flow cytometry. Compare results to 12-month Relapse-Free Survival rate using statistical analysis.
Time Frame: 12-months
Reporting Status: Not Posted

25. Secondary Outcome: Ratio of T-cell Subpopulations
Description: Ratio of t-cell subpopulations utilizing IHC staining and flow cytometry. Compare results to 12-month Relapse-Free Survival rate using statistical analysis.
Time Frame: 12-months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Intravesical Gemcitabine/Docetaxel
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 2/26
Other Adverse Events (participants affected / at risk) | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravesical Gemcitabine/Docetaxel (N=26)
Urinary tract infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravesical Gemcitabine/Docetaxel (N=26)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 3 (3)
Blurred vision (Eye disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 4 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Eye disorders - Other, Meibomian gland dysfunction (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 9 (9)
Fever (General disorders) | 2 (2)
Gait disturbance (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 8 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 4 (4)
Insomnia (Psychiatric disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Metabolism and nutrition disorders - Other, Type II Diabetes (Metabolism and nutrition disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5)
Nervous system disorders - Other, Parkinson's disease (Nervous system disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Renal and urinary disorders - Other, lower urinary tract symptoms (Renal and urinary disorders) | 3 (3)
Renal and urinary disorders - Other, docetaxel retention (Renal and urinary disorders) | 1 (1)
Reproductive system and breast disorders - Other, right breast tenderness (Reproductive system and breast disorders) | 1 (1)
Retinopathy (Eye disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Urinary tract infection (Renal and urinary disorders) | 5 (6)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT04386746/Prot_SAP_000.pdf